CLINICAL TRIAL: NCT03713723
Title: Cardiac Output Monitoring in Patients Undergoing In Vitro Fertilization by Noninvasive Cardiac Impendence: A Prospective Observational Study
Brief Title: Cardiac Output Monitoring in IVF Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 172-17
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2018-10

CONDITIONS: Fertilization in Vitro

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Patients undergoing IVF treatment with hemodynamic monitoring: Fifty health women aged 18-45 undergoing their first, second or third cycle of IVF treatment will be monitored with the non invasive NICaS bioimpedance
  Interventions: Device: NICaS bioimpedance system

INTERVENTIONS:
Device: NICaS bioimpedance system — NICaS is a bioimpedance system focusing on noninvasive assessment and monitoring of cardiovascular, respiratory, and fluid parameters.Cardiovascular monitoring will be carried out using non-invasive NICAS cardiac impedance cardiography by the use of two electrodes stickers which are pasted on the wrists for 6 minutes

SUMMARY:
In this study we aim to evaluate hemodynamic effects of IVF treatment, with the use of the non invasive NICaS bioimpendence monitor.

Our study's primary end point is to evaluate the hemodynamic profile with the use of NICaS whole body impedance cardiography that occur throughout the IVF cycle in patients undergoing controlled ovarian stimulation during IVF treatment.

Secondary endpoints include:

Women will be asked to grade their pain score and level of anxiety by the use of the visual analogue score elicited throughout the study observation points, in order to examine whether pain scores and anxiety levels correlate with the hemodynamic changes throughout an IVF treatment cycle.

DETAILED DESCRIPTION:
This is a prospective, observational, single center study which will be conducted at the Rabin Medical Center (Beilinson Campus), Petach Tikva, Israel, a tertiary university hospital. Fifty healthy woman (≤45 years old) undergoing IVF treatment will be enrolled following filling out an informed consent form.

Study procedure:

Women will be recruited in the IVF department upon consulting with the fertility specialist. Following signed informed consent, patients' blood pressure will be measured using a non-invasive upper arm blood pressure. Cardiovascular monitoring will be carried out using non-invasive NICAS cardiac impedance cardiography by the use of two electrodes stickers which are pasted on the wrists for 6 minutes.

Monitoring will be performed on:

1. 1-3rd day of the menstrual cycle prior to treatment with gonadotropins
2. On the day of ovulation triggering
3. On the day of ovum pickup prior to their entrance to the operating theater.
4. On the day of embryo transfer.

IVF Protocol:

The antagonist protocol consists of daily gonadotropin stimulation from day 3 or 4 of menstruation. In addition, once the leading follicle reached 13-14 mm, daily injections of Cetrotide 0.25 mg (Serono, Switzerland) or Orgalutran 0.25 mg (N.V. Organon, the Netherlands) are given and until the day of hCG (Ovitrelle, Serono, Switzerland) injection. Gonadotropin stimulation will consist of recombinant FSH (Gonal F, Serono, Postfach, Switzerland; or Puregon, N.V. Organon, Oss, The Netherlands), alone or in combination with urinary gonadotropins (Menopur, Ferring, Kiel, Germany). During treatment, the ovarian response will be monitored by serial vaginal ultrasound measurements of follicular growth and serum E2 level every 1-3 days, starting on the fourth or fifth day of stimulation, gonadotropin dosage will be adjusted accordingly. When at least 3 follicles reached at least 17 millimeters, hCG is injected and thirty six hours after hCG injection, follicles will be aspirated in the operating room.

Data Collection:

Recorded data will include:

* Cardiac Output and its derivate including: systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), heart rate (HR), stroke volume (SV), cardiac output (CO) and total peripheral resistance (TPR).
* Demographic and obstetric age, weight, height, current hemoglobin, comorbidities, regular medication and other obstetric data.

Data Handling Data collection for all participants in the study will be done anonymously. All hemodynamic data collected will be done by a trained member of the research team. All collected data will be coded and recorded on the eCRF NICaS monitor, and will be accessible only to a member of the research team.

Study duration:

The study duration for each participant will be throughout the IVF cycle of treatment approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

Women above 18-45 undergoing their first, second or third cycle of IVF treatment in Beilinson Hospital following obtaining written informed consents forums with the ability to comply with the study requirements will be included in our study.

Exclusion Criteria:

* Women under age 18
* Women with polycystic ovarian syndrome
* Women with cardiomyopathy
* Women with history of chronic hypertension
* Women with a congenital heart disease
* Women who are not able to comply with study requirements and can't sign an informed consent forum.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: This is a prospective, observational, single center study which will be conducted at the Rabin Medical Center (Beilinson Campus), Petach Tikva, Israel, a tertiary university hospital. Fifty healthy woman (≤45 years old) undergoing IVF treatment will be enrolled following filling out an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac output measurement with the use of non-invasive NICAS hemodynamic monitor | On the day of ovum pickup prior to their entrance to the operating theater.

SECONDARY OUTCOMES:
Cardiac output measurement with the use of non-invasive NICAS hemodynamic monitor | 1-3rd day of the menstrual cycle prior to treatment with gonadotropins

CONTACTS AND LOCATIONS:
Locations (1):
- Beilinson hospital, Petach Tikvah, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harnett MJ, Bhavani-Shankar K, Datta S, Tsen LC. In vitro fertilization-induced alterations in coagulation and fibrinolysis as measured by thromboelastography. Anesth Analg. 2002 Oct;95(4):1063-6, table of contents. doi: 10.1097/00000539-200210000-00050. PMID 12351295
- [Background] Orbach-Zinger S, Eidelman LA, Lutsker A, Oron G, Fisch B, Ben-Haroush A. The effect of in vitro fertilization on coagulation parameters as measured by thromboelastogram. Eur J Obstet Gynecol Reprod Biol. 2016 Jun;201:118-20. doi: 10.1016/j.ejogrb.2016.04.010. Epub 2016 Apr 11. PMID 27092869
- [Background] Manau D, Fabregues F, Arroyo V, Jimenez W, Vanrell JA, Balasch J. Hemodynamic changes induced by urinary human chorionic gonadotropin and recombinant luteinizing hormone used for inducing final follicular maturation and luteinization. Fertil Steril. 2002 Dec;78(6):1261-7. doi: 10.1016/s0015-0282(02)04394-7. PMID 12477522
- [Background] Barbieri RL, Hornstein MD. Assisted reproduction-in vitro fertilization success is improved by ovarian stimulation with exogenous gonadotropins and pituitary suppression with gonadotropin-releasing hormone analogues. Endocr Rev. 1999 Jun;20(3):249-52. doi: 10.1210/edrv.20.3.0363. No abstract available. PMID 10368770
- [Background] Magnani B, Tsen L, Datta S, Bader A. In vitro fertilization. Do short-term changes in estrogen levels produce increased fibrinolysis? Am J Clin Pathol. 1999 Oct;112(4):485-91. doi: 10.1093/ajcp/112.4.485. PMID 10510672
- [Background] Aurousseau MH, Samama MM, Belhassen A, Herve F, Hugues JN. Risk of thromboembolism in relation to an in-vitro fertilization programme: three case reports. Hum Reprod. 1995 Jan;10(1):94-7. doi: 10.1093/humrep/10.1.94. PMID 7745079
- [Background] Westerlund E, Antovic A, Hovatta O, Eberg KP, Blomback M, Wallen H, Henriksson P. Changes in von Willebrand factor and ADAMTS13 during IVF. Blood Coagul Fibrinolysis. 2011 Mar;22(2):127-31. doi: 10.1097/MBC.0b013e32834363ea. PMID 21192251
- [Background] Biron C, Galtier-Dereure F, Rabesandratana H, Bernard I, Aguilar-Martinez P, Schved JF, Hedon B. Hemostasis parameters during ovarian stimulation for in vitro fertilization: results of a prospective study. Fertil Steril. 1997 Jan;67(1):104-9. doi: 10.1016/s0015-0282(97)81864-x. PMID 8986692
- [Background] Bremme K, Wramsby H, Andersson O, Wallin M, Blomback M. Do lowered factor VII levels at extremely high endogenous oestradiol levels protect against thrombin formation? Blood Coagul Fibrinolysis. 1994 Apr;5(2):205-10. doi: 10.1097/00001721-199404000-00008. PMID 8054452
- [Background] Curvers J, Nap AW, Thomassen MC, Nienhuis SJ, Hamulyak K, Evers JL, Tans G, Rosing J. Effect of in vitro fertilization treatment and subsequent pregnancy on the protein C pathway. Br J Haematol. 2001 Nov;115(2):400-7. doi: 10.1046/j.1365-2141.2001.03118.x. PMID 11703342
- [Background] Chan WS, Dixon ME. The "ART" of thromboembolism: a review of assisted reproductive technology and thromboembolic complications. Thromb Res. 2008;121(6):713-26. doi: 10.1016/j.thromres.2007.05.023. Epub 2007 Jul 30. PMID 17659766
- [Background] Ogawa S, Minakami H, Araki S, Ohno T, Motoyama M, Shibahara H, Sato I. A rise of the serum level of von Willebrand factor occurs before clinical manifestation of the severe form of ovarian hyperstimulation syndrome. J Assist Reprod Genet. 2001 Feb;18(2):114-9. doi: 10.1023/a:1026590910462. PMID 11285978
- [Background] Richter ON, Kubler K, Schmolling J, Kupka M, Reinsberg J, Ulrich U, van der Ven H, Wardelmann E, van der Ven K. Oxytocin receptor gene expression of estrogen-stimulated human myometrium in extracorporeally perfused non-pregnant uteri. Mol Hum Reprod. 2004 May;10(5):339-46. doi: 10.1093/molehr/gah039. Epub 2004 Mar 25. PMID 15044599
- [Background] Liedman R, Hansson SR, Howe D, Igidbashian S, McLeod A, Russell RJ, Akerlund M. Reproductive hormones in plasma over the menstrual cycle in primary dysmenorrhea compared with healthy subjects. Gynecol Endocrinol. 2008 Sep;24(9):508-13. doi: 10.1080/09513590802306218. PMID 18958771
- [Background] Gizzo S, Noventa M, Quaranta M, Vitagliano A, Esposito F, Andrisani A, Venturella R, Alviggi C, Plebani M, Gangemi M, Nardelli GB, D'Antona D. The Potential Role of GnRH Agonists and Antagonists in Inducing Thyroid Physiopathological Changes During IVF. Reprod Sci. 2016 Apr;23(4):515-23. doi: 10.1177/1933719115608000. Epub 2015 Oct 6. PMID 26445999
- [Background] Mintziori G, Goulis DG, Toulis KA, Venetis CA, Kolibianakis EM, Tarlatzis BC. Thyroid function during ovarian stimulation: a systematic review. Fertil Steril. 2011 Sep;96(3):780-5. doi: 10.1016/j.fertnstert.2011.06.020. Epub 2011 Jul 13. PMID 21742326
- [Background] Benaglia L, Busnelli A, Somigliana E, Leonardi M, Vannucchi G, De Leo S, Fugazzola L, Ragni G, Fedele L. Incidence of elevation of serum thyroid-stimulating hormone during controlled ovarian hyperstimulation for in vitro fertilization. Eur J Obstet Gynecol Reprod Biol. 2014 Feb;173:53-7. doi: 10.1016/j.ejogrb.2013.11.003. Epub 2013 Nov 9. PMID 24332278
- [Background] Persson M, Ekerfelt C, Jablonowska B, Jonsson Y, Ernerudh J, Jenmalm MC, Berg G. Immunological status in patients undergoing in vitro fertilisation: responses to hormone treatment and relationship to outcome. J Reprod Immunol. 2012 Dec;96(1-2):58-67. doi: 10.1016/j.jri.2012.07.005. Epub 2012 Sep 13. PMID 22981121
- [Background] Liang PY, Yin B, Cai J, Hu XD, Song C, Wu TH, Zhao J, Li GG, Zeng Y. Increased circulating Th1/Th2 ratios but not other lymphocyte subsets during controlled ovarian stimulation are linked to subsequent implantation failure after transfer of in vitro fertilized embryos. Am J Reprod Immunol. 2015 Jan;73(1):12-21. doi: 10.1111/aji.12320. Epub 2014 Sep 15. PMID 25220906
- [Background] Kalu E, Bhaskaran S, Thum MY, Vishwanatha R, Croucher C, Sherriff E, Ford B, Bansal AS. Serial estimation of Th1:th2 cytokines profile in women undergoing in-vitro fertilization-embryo transfer. Am J Reprod Immunol. 2008 Mar;59(3):206-11. doi: 10.1111/j.1600-0897.2007.00565.x. PMID 18275514
- [Background] Salmassi A, Schmutzler AG, Schaefer S, Koch K, Hedderich J, Jonat W, Mettler L. Is granulocyte colony-stimulating factor level predictive for human IVF outcome? Hum Reprod. 2005 Sep;20(9):2434-40. doi: 10.1093/humrep/dei071. Epub 2005 May 12. PMID 15890733
- [Background] Salmassi A, Mettler L, Jonat W, Buck S, Koch K, Schmutzler AG. Circulating level of macrophage colony-stimulating factor can be predictive for human in vitro fertilization outcome. Fertil Steril. 2010 Jan;93(1):116-23. doi: 10.1016/j.fertnstert.2008.09.083. Epub 2008 Nov 8. PMID 18996518
- [Background] Wu MY, Chen HF, Chen SU, Chao KH, Yang YS, Ho HN. Increase in the production of interleukin-10 early after implantation is related to the success of pregnancy. Am J Reprod Immunol. 2001 Dec;46(6):386-92. doi: 10.1034/j.1600-0897.2001.d01-29.x. PMID 11775007
- [Background] Manau D, Balasch J, Arroyo V, Jimenez W, Fabregues F, Casamitjana R, Creus M, Vanrell JA. Circulatory dysfunction in asymptomatic in vitro fertilization patients. Relationship with hyperestrogenemia and activity of endogenous vasodilators. J Clin Endocrinol Metab. 1998 May;83(5):1489-93. doi: 10.1210/jcem.83.5.4796. PMID 9589644
- [Background] Manau D, Arroyo V, Jimenez W, Fabregues F, Vanrell JA, Balasch J. Chronology of hemodynamic changes in asymptomatic in vitro fertilization patients and relationship with ovarian steroids and cytokines. Fertil Steril. 2002 Jun;77(6):1178-83. doi: 10.1016/s0015-0282(02)03116-3. PMID 12057725
- [Background] Armstrong S, Fernando R, Columb M. Minimally- and non-invasive assessment of maternal cardiac output: go with the flow! Int J Obstet Anesth. 2011 Oct;20(4):330-40. doi: 10.1016/j.ijoa.2011.07.006. Epub 2011 Sep 16. PMID 21925868
- [Background] Cotter G, Moshkovitz Y, Kaluski E, Cohen AJ, Miller H, Goor D, Vered Z. Accurate, noninvasive continuous monitoring of cardiac output by whole-body electrical bioimpedance. Chest. 2004 Apr;125(4):1431-40. doi: 10.1378/chest.125.4.1431. PMID 15078756
- [Background] Taniguchi Y, Emoto N, Miyagawa K, Nakayama K, Kinutani H, Tanaka H, Shinke T, Hirata K. Noninvasive and simple assessment of cardiac output and pulmonary vascular resistance with whole-body impedance cardiography is useful for monitoring patients with pulmonary hypertension. Circ J. 2013;77(9):2383-9. doi: 10.1253/circj.cj-13-0172. Epub 2013 Jun 12. PMID 23759655